CLINICAL TRIAL: NCT01523873
Title: Observational Post-marketing Study on the Safety and Efficacy of Dotarem® (SECURE Study)
Status: Completed | Type: Observational
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: DGD-55-001
Record Dates: First submitted 2012-01-26; First posted 2012-02-01 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: General Safety Profile of DOTAREM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The main purpose of this study is to prospectively assess the general safety profile of Dotarem

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for a Dotarem®-enhanced MRI

Exclusion Criteria:

* patient with a contra-indication to MR examination
* patient with a contra-indication to Dotarem® injection as per local SPC

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients scheduled for a Dotarem®-enhanced MRI over a one year period at each participating radiological site
Sampling Method: Non-Probability Sample
Enrollment: 35921 (Actual)
Dates: Start 2008-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Diagnosticum Gersthof, Vienna, Austria
- Shanghai Pulmonary Hospital, Shanghai, China
- Hôpital Necker, Paris, France
- Universitätskliniken, Cologne, Germany
- Bombay Hospital Institute of Medical Sciences, Mumbai, India
- Ospedale Policlinico Giambattista Rossi, Verona, Italy
- Tabouk Military Hospital, Tabuk, Saudi Arabia
- Complexo Hospitalario Xeral-Calde, Lugo, Spain
- Hull Royal Infirmary, Hull, United Kingdom

REFERENCES:
- [Derived] Heshmatzadeh Behzadi A, McDonald J. Gadolinium-based contrast agents for imaging of the central nervous system: A multicenter European prospective study. Medicine (Baltimore). 2022 Aug 26;101(34):e30163. doi: 10.1097/MD.0000000000030163. PMID 36042629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for a Dotarem-enhanced MRI were recruited in 118 active centers in 10 countries from November 2008 to June 2013.
Groups:
- All Included Patients: All patients scheduled for a Dotarem-enhanced MRI with appropriate consent, prospectively enrolled in the study and having reliable data reported.
Period: Overall Study
Arm/Group | All Included Patients
Started | 35921
Administered With Dotarem | 35474
Completed | 35499
Not Completed | 422
Not completed — Protocol Violation | 422

BASELINE CHARACTERISTICS:
Arm/Group | All Included Patients
Number analyzed (Participants) | 35499
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data were missing for 144 patients.
  years
    number analyzed (Participants) | 35355
    (all) | 49.5 (17.9)
Age, Customized [Number; unit: participants] — Population: Data were missing for 75 patients.
  participants
    <18 years: number analyzed (Participants) | 35424
    <18 years | 1631
    from 18 to 64 years: number analyzed (Participants) | 35424
    from 18 to 64 years | 26058
    ≥65 years: number analyzed (Participants) | 35424
    ≥65 years | 7735
Gender [Count of Participants; unit: Participants] — Population: Data were missing for 41 patients.
  Participants
    number analyzed (Participants) | 35458
    Female | 18838
    Male | 16620
Region of Enrollment [Number; unit: participants]
  France | 7692
  Argentina | 43
  Austria | 703
  China | 7064
  Germany | 9988
  India | 6803
  Italy | 328
  Saudi Arabia | 372
  Spain | 1039
  United Kingdom | 1467

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: Adverse Events were notified and described.
Time Frame: During the time of usual follow-up post Dotarem administration (from less than 30 min to 1 hour after magnetic resonance examination).
Measure: Number; unit: Adverse Events
Groups:
- Safety Population: Safety Population included All Included Patients administered with Dotarem.
Arm/Group | Safety Population
Number analyzed (Participants) | 35474
Adverse Events | 70

2. Secondary Outcome: Nephrogenic Systemic Fibrosis Incidence
Description: For any patient identified with moderate to severe impaired renal function at the time of inclusion, a specific safety follow-up was performed in order to detect any suspicion of Nephrogenic Systemic Fibrosis.
Time Frame: Follow-up of at least 3 months after magnetic resonance examination
Population: Patients of the Safety Population with moderate to severe impaired renal function.
Measure: Number; unit: participants
Groups:
- Patients With Moderate to Severe Impaired Renal Function: Patients identified with moderate to severe impaired renal function at the time of inclusion (i.e. estimated Glomerular Filtration Rate (eGFR) or estimated creatinine clearance (eCrCl) <60 ml/min (1.73 m2))
Arm/Group | Patients With Moderate to Severe Impaired Renal Function
Number analyzed (Participants) | 514
participants | 0

3. Secondary Outcome: Image Quality
Description: Image quality was assessed by the radiologist using a scale with five classes: very poor, poor, fair, good and very good.
Time Frame: Up to 1 hour (as the duration of usual follow-up post Dotarem administration was from less than 30 min to 1 hour)
Population: Data were missing for 164 patients.
Measure: Number; unit: participants
Groups:
- Efficacy Population: Efficacy Population included all patients administered with Dotarem who have been imaged and have had a valid diagnostic assessment.
Arm/Group | Efficacy Population
Number analyzed (Participants) | 34572
participants
  very poor | 6
  poor | 52
  fair | 341
  good | 10268
  very good | 23741

4. Secondary Outcome: Diagnostic Quality
Description: Diagnostic quality was assessed by the radiologist by answering the question "could you come to a diagnostic ?" (answer : yes or no).
Time Frame: Up to 1 hour (as the duration of usual follow-up post Dotarem administration was from less than 30 min to 1 hour)
Population: Data were missing for 308 patients.
Measure: Number; unit: participants
Arm/Group | Efficacy Population
Number analyzed (Participants) | 34572
participants
  No | 343
  Yes | 33921

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded during the time of usual follow-up post Dotarem administration (from less than 30 min to 1 hour after magnetic resonance examination).
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 9/35474
Other Adverse Events (participants affected / at risk) | 35/35474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=35474)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Adverse event (General disorders) | 2 (2)
Death (General disorders) | 2 (2)
General physic health deterioration (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Candida sepsis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=35474)
Vomiting (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 7 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Extravasation (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site extravasation (General disorders) | 1 (1)
Injection site warmth (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Clonus (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No